CLINICAL TRIAL: NCT06623422
Title: A Phase 3 Randomized Double-blind Study of Adjuvant Pembrolizumab With or Without V940 in Participants With Resectable Stage II to IIIB (N2) NSCLC Not Achieving pCR After Receiving Neoadjuvant Pembrolizumab With Platinum-based Doublet Chemotherapy (INTerpath-009)
Brief Title: A Study of Pembrolizumab (MK-3475) With or Without Intismeran Autogene (V940) in Participants With Non-small Cell Lung Cancer (V940-009/INTerpath-009)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V940-009; 2023-506327-29-00 (Registry Identifier: EU CT); U1111-1293-5814 (Registry Identifier: UTN); INTerpath-009 (Other: MSD); jRCT2061240105 (Registry Identifier: jRCT)
Record Dates: First submitted 2024-09-05; First posted 2024-10-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2); Individualized neoantigen therapy (INT)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Cisplatin; Carboplatin; Pemetrexed; Gemcitabine; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Intismeran autogene (Experimental): For neoadjuvant treatment, participants will receive pembrolizumab 200 mg via intravenous (IV) infusion every 3-week cycle for up to 4 cycles PLUS background chemotherapy via IV infusion (cisplatin 75 mg/m^2 or carboplatin area under the curve [AUC] 5 or 6 mg/mL/min, pemetrexed 500 mg/m^2, gemcitabine 1000 mg/m^2, paclitaxel 175 mg/m^2 or 200 mg/m^2 given at a dose and combination per investigator's choice) every 3-week cycle for up to 4 cycles (total neoadjuvant treatment duration of up to ~12 weeks). After surgical resection, for adjuvant treatment, participants will receive pembrolizumab 400 mg via IV infusion every 6-week cycle for up to 7 cycles PLUS intismeran autogene 1 mg via intramuscular (IM) injection every 3 weeks for up to 9 doses (total adjuvant treatment duration of up to ~42 weeks).
  Interventions: Biological: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: Gemcitabine; Drug: Paclitaxel; Biological: Intismeran autogene
- Pembrolizumab + Placebo (Active Comparator): For neoadjuvant treatment, participants will receive pembrolizumab 200 mg via IV infusion every 3-week cycle for up to 4 cycles PLUS background chemotherapy via IV infusion (cisplatin 75 mg/m^2 or carboplatin AUC 5 or 6 mg/mL/min, pemetrexed 500 mg/m^2, gemcitabine 1000 mg/m^2, paclitaxel 175 mg/m^2 or 200 mg/m^2 given at a dose and combination per investigator's choice) every 3-week cycle for up to 4 cycles (total neoadjuvant treatment duration of up to ~12 weeks). After surgical resection, for adjuvant treatment, participants will receive pembrolizumab 400 mg via IV infusion every 6-week cycle for up to 7 cycles PLUS matching placebo via IM injection every 3 weeks for up to 9 doses (total adjuvant treatment duration of up to ~42 weeks).
  Interventions: Biological: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: Gemcitabine; Drug: Paclitaxel; Other: Placebo

INTERVENTIONS:
Biological: Pembrolizumab — IV Infusion
  Other Names: MK-3475; KEYTRUDA®
Drug: Cisplatin — IV infusion
  Other Names: Platinol®; Platinol®-AQ
Drug: Carboplatin — IV infusion
  Other Names: Paraplatin®
Drug: Pemetrexed — IV infusion
  Other Names: Alimta®
Drug: Gemcitabine — IV infusion
  Other Names: Gemzar
Drug: Paclitaxel — IV infusion
  Other Names: Taxol®; Onxol®
Biological: Intismeran autogene — IM injection
  Other Names: mRNA-4157; V940
  Arms: Pembrolizumab + Intismeran autogene
Other: Placebo — IM injection
  Arms: Pembrolizumab + Placebo

SUMMARY:
The goal of this study is to learn if people who receive intismeran autogene and pembrolizumab after surgery are cancer-free longer than people who receive placebo and pembrolizumab. Researchers want to know if giving intismeran autogene and pembrolizumab after surgery can help prevent the cancer from coming back in people with non-small cell lung cancer (NSCLC) whose tumors did not respond completely to treatment before surgery (neoadjuvant treatment).

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has histologically/cytologically confirmed diagnosis of previously untreated and pathologically confirmed resectable Stage II, IIIA, or IIIB (N2) non-small cell lung cancer (NSCLC) [American Joint Committee on Cancer (AJCC) 8th Edition]
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days before the first dose of study intervention
* Participants who have not achieved a pathological complete response (pCR) following completion of neoadjuvant chemotherapy and pembrolizumab followed by surgery will be eligible
* Confirmation that epidermal growth factor receptor (EGFR)-directed therapy is not indicated as primary therapy (documentation of absence of tumor-activating EGFR mutations [eg, DEL19 or L858R])
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on anti-retroviral therapy (ART)
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization
* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Diagnosis of SCLC or, for mixed tumors, presence of small cell elements, or has a neuroendocrine tumor with large-cell components, or a sarcomatoid carcinoma, or a pancoast tumor
* Documentation by local test report indicating presence of anaplastic lymphoma kinase (ALK) gene rearrangements
* Received prior neoadjuvant therapy for their current NSCLC diagnosis
* Received prior therapy with an anti-programmed cell death 1 (PD-1), anti-programmed cell death ligand 1 (PD-L1), or anti-programmed cell-death ligand 2 (PD-L2) agent, or with an agent directed to another stimulatory or coinhibitory T-cell receptor (eg, cytotoxic T-lymphocyte-associated protein [CTLA-4], OX-40, CD137)
* Received prior systemic anticancer therapy including investigational agents other than what is specified in this protocol
* Received prior treatment with a cancer vaccine
* Received prior radiotherapy within 2 weeks of start of study intervention, or has radiation-related toxicities, requiring corticosteroids
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2033-05-16 (Estimated); Study Completion 2038-01-26 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | Up to ~97 months
  DFS is defined as the time from randomization to any recurrence (local, locoregional, regional or distant), occurrence of new primary NSCLC, as assessed by the investigator, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to ~129 months
  OS is defined as the time from randomization to death due to any cause.
Distant Metastasis-Free Survival (DMFS) | Up to ~129 months
  DMFS is defined as the time from randomization to the first diagnosis of a distant metastasis as assessed by the investigator, or death due to any cause, whichever occurs first. Distant metastasis refers to cancer that has spread from the original (primary) tumor and beyond local tissues and lymph nodes to distant organs or distant lymph nodes.
Disease-Free Survival 2 (DFS2) | Up to ~129 months
  DFS2 is defined as the time from randomization to subsequent recurrence or disease progression after initiation of next-line anticancer therapy as assessed by the investigator, or death due to any cause, whichever occurs first.
Lung Cancer Specific Survival (LCSS) | Up to ~129 months
  LCSS is defined as the time from randomization to death due to lung cancer specifically as assessed by the investigator.
Change from Baseline in the European Organization for Research and Treatment of Cancer (EORTC)-Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status/Quality of Life (Items 29 and 30) | Baseline and up to ~129 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" will be scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores will be standardized, so that scores range from 0 to 100. Higher scores indicate a better overall health status. The change from baseline in global health status/quality of life (EORTC QLQ-C30 Items 29 and 30) combined score will be presented.
Change from Baseline in the EORTC QLQ-C30 Physical Functioning (Items 1-5) | Baseline and up to ~129 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to 5 questions about their physical functioning will be scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores will be standardized, so that scores range from 0 to 100. Higher scores indicate a worse level of physical functioning. The change from baseline in physical functioning (EORTC QLQ-C30 Items 1-5) combined score will be presented.
Change from Baseline in the EORTC QLQ-C30 Role Functioning (Items 6 and 7) | Baseline and up to ~129 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "Were you limited in doing either your work or other daily activities during the past week?" and " Were you limited in pursuing your hobbies or other leisure time activities during the past week?" will be scored on a 4-point scale (1=Not at All to 4=Very Much). Higher scores indicate a worse level of role functioning. Change from baseline in the role functioning (EORTC QLQ-C30 Items 6 and 7) combined score will be presented.
Number of participants with ≥1 adverse event (AE) | Up to ~129 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants discontinuing from study therapy due to AE(s) | Up to ~129 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (219):
- United States (46):
  - Banner MD Anderson Cancer Center ( Site 0181), Gilbert, Arizona
  - Providence St. Jude Medical Center ( Site 0106), Fullerton, California
  - VA Long Beach Healthcare System ( Site 0199), Long Beach, California
  - USC Norris Comprehensive Cancer Center ( Site 0205), Los Angeles, California
  - UCSF Medical Center at Mission Bay ( Site 0178), San Francisco, California
  - University of Colorado Anschutz Medical Campus ( Site 0151), Aurora, Colorado
  - UCHealth Memorial Hospital Central ( Site 0125), Colorado Springs, Colorado
  - Banner MD Anderson Cancer Center at North Colorado Medical Center ( Site 0207), Greeley, Colorado
  - Centura Health - St. Anthony North Health Campus ( Site 0189), Westminster, Colorado
  - Yale University School of Medicine ( Site 0201), New Haven, Connecticut
  - Eastern CT Hematology & Oncology Associates ( Site 0202), Norwich, Connecticut
  - The Oncology Institute of Hope and Innovation - Fort Lauderdale ( Site 0156), Fort Lauderdale, Florida
  - Beacon Cancer Care ( Site 0127), Post Falls, Idaho
  - The University of Chicago Medical Center ( Site 0118), Chicago, Illinois
  - Maryland Oncology Hematology (MOH) ( Site 8102), Rockville, Maryland
  - Massachusetts General Hospital ( Site 0136), Boston, Massachusetts
  - Dana Farber Cancer Hospital ( Site 0155), Boston, Massachusetts
  - Ellis Fischel Cancer Center ( Site 0133), Columbia, Missouri
  - Lake Regional Hospital-Cancer Center ( Site 0123), Osage Beach, Missouri
  - Roswell Park Cancer Institute ( Site 0184), Buffalo, New York
  - Hematology-Oncology Associates of CNY ( Site 0164), East Syracuse, New York
  - The Blavatnik Family- Chelsea Medical Center at Mount Sinai ( Site 0216), New York, New York
  - Icahn School of Medicine at Mount Sinai ( Site 0116), New York, New York
  - Memorial Sloan Kettering Cancer Center ( Site 0137), New York, New York
  - SUNY Upstate Cancer Center ( Site 0140), Syracuse, New York
  - Montefiore Medical Center ( Site 0160), The Bronx, New York
  - Westchester Medical Center ( Site 0196), Valhalla, New York
  - Novant Health Weisiger Cancer Insititute ( Site 0266), Charlotte, North Carolina
  - Novant Health Forsyth Medical Center ( Site 0166), Winston-Salem, North Carolina
  - University of Cincinnati Medical Center ( Site 0119), Cincinnati, Ohio
  - St. Lukes Hospital and Health Network ( Site 0186), Bethlehem, Pennsylvania
  - Thompson Cancer Survival Center ( Site 0168), Knoxville, Tennessee
  - Elliston Place Medical Oncology & Hematology ( Site 0215), Nashville, Tennessee
  - Texas Oncology - DFW ( Site 8103), Dallas, Texas
  - UT Southwestern Medical Center ( Site 0190), Dallas, Texas
  - Houston Methodist Cancer Center ( Site 0191), Houston, Texas
  - MD Anderson Cancer Center ( Site 0150), Houston, Texas
  - Memorial Hermann Cancer Center ( Site 0172), Houston, Texas
  - Michael E. DeBakey VA Medical Center ( Site 0197), Houston, Texas
  - O'Quinn Medical Tower at McNair Campus ( Site 0131), Houston, Texas
  - The University of Texas Health Science Center at Tyler dba UT Health East Texas HOPE Cancer Center ( Site 0148), Tyler, Texas
  - Virginia Cancer Specialists ( Site 0167), Fairfax, Virginia
  - Virginia Oncology Associates (VOA) ( Site 8101), Norfolk, Virginia
  - VCU Health Adult Outpatient Pavillion ( Site 0193), Richmond, Virginia
  - Swedish Cancer Institute ( Site 0143), Seattle, Washington
  - Virginia Mason Franciscan Health - St. Michael Cancer Center ( Site 0192), Silverdale, Washington
- Argentina (6):
  - CEMIC ( Site 2454), Caba., Buenos Aires
  - Hospital Italiano de Buenos Aires-Clinical Oncology ( Site 2459), Ciudad Autonoma de Buenos Aires., Buenos Aires
  - Fundacion Intecnus ( Site 2456), Bariloche, Río Negro Province
  - Centro Médico IPAM ( Site 2452), Rosario, Santa Fe Province
  - Instituto Medico Especializado Alexander Fleming ( Site 2457), Buenos Aires
  - Instituto Oncologico de Cordoba -IONC ( Site 2455), Córdoba
- Australia (5):
  - Calvary Mater Newcastle ( Site 2106), Waratah, New South Wales
  - Tasman Oncology Research ( Site 2104), Southport, Queensland
  - Princess Alexandra Hospital ( Site 2102), Wooloongabba, Queensland
  - Grampians Health ( Site 2101), Ballarat, Victoria
  - One Clinical Research ( Site 2103), Nedlands, Western Australia
- Belgium (3):
  - Cliniques Universitaires Saint-Luc ( Site 1203), Brussels, Bruxelles-Capitale, Region de
  - Jessa Ziekenhuis ( Site 1204), Hasselt, Limburg
  - UZ Gent ( Site 1201), Ghent, Oost-Vlaanderen
- Brazil (9):
  - CRIO - CENTRO REGIONAL INTEGRADO DE ONCOLOGIA ( Site 2502), Fortaleza, Ceará
  - Liga Norte Riograndense Contra o Cancer ( Site 2513), Natal, Rio Grande do Norte
  - Hospital Tacchini ( Site 2506), Bento Gonçalves, Rio Grande do Sul
  - Hospital de Clínicas de Passo Fundo ( Site 2504), Passo Fundo, Rio Grande do Sul
  - Hospital Moinhos de Vento ( Site 2510), Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora Da Conceicao ( Site 2512), Porto Alegre, Rio Grande do Sul
  - Instituto de Oncologia Saint Gallen ( Site 2507), Santa Cruz do Sul, Rio Grande do Sul
  - Hospital de Amor - Barretos ( Site 2511), Barretos, São Paulo
  - Instituto Nacional de Câncer - INCA ( Site 2501), Rio de Janeiro
- Bulgaria (2):
  - MBAL Uni Hospital ( Site 1253), Panagyurishte, Pazardzhik
  - MHAT - Heart and Brain ( Site 1252), Pleven
- Canada (7):
  - Queen Elizabeth II Health Sciences Centre ( Site 1101), Halifax, Nova Scotia
  - Hamilton Health Sciences - Juravinski Site ( Site 1104), Hamilton, Ontario
  - Kingston Health Sciences Centre-Kingston General Hospital Site ( Site 1105), Kingston, Ontario
  - Lakeridge Health ( Site 1107), Oshawa, Ontario
  - Sunnybrook Research Institute ( Site 1106), Toronto, Ontario
  - McGill University Health Centre ( Site 1103), Montreal, Quebec
  - IUCPQ ( Site 1112), Québec, Quebec
- Chile (5):
  - Orlandi Oncologia ( Site 2555), Santiago, Region M. de Santiago
  - FALP ( Site 2551), Santiago, Region M. de Santiago
  - Clínica RedSalud Vitacura ( Site 2556), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 2552), Santiago, Region M. de Santiago
  - ONCOCENTRO APYS ( Site 2554), Viña del Mar, Región de Valparaíso
- Colombia (6):
  - FUNDACION CTIC CENTRO DE TRATAMIENTO E INVESTIGACION SOBRE CANCER LUIS CARLOS SARMIENTO ANGULO ( Site 2603), Bogotá, Bogota D.C.
  - Hospital Universitario San Ignacio ( Site 2610), Bogotá, Bogota D.C.
  - Clinica Colsanitas S.A, Sede Clínica Universitaria Colombia ( Site 2604), Bogotá, Bogota D.C.
  - IMAT S.A.S ( Site 2602), Montería, Departamento de Córdoba
  - Oncologos del Occidente ( Site 2608), Pereira, Risaralda Department
  - Fundacion Valle del Lili- CIC ( Site 2601), Cali, Valle del Cauca Department
- Finland (2):
  - Oulun yliopistollinen sairaala ( Site 1301), Oulu, Northern Savonia
  - Turku University Hospital ( Site 1303), Turku, Southwest Finland
- France (6):
  - Centre Hospitalier Régional Universitaire de Tours - Hôpital Bretonneau ( Site 1354), Tours, Centre-Val de Loire
  - CHU Besançon ( Site 1358), Besançon, Franche-Comte
  - Institut De Cancerologie De L Ouest ( Site 1357), Saint-Herblain, Loire-Atlantique
  - Institut Cœur Poumon -CHU Lille ( Site 1352), Lille, Nord
  - CENTRE LEON BERARD ( Site 1351), Lyon, Rhone
  - Gustave Roussy ( Site 1353), Villejuif, Île-de-France Region
- Germany (7):
  - Robert-Bosch-Krankenhaus ( Site 1401), Stuttgart, Baden-Wurttemberg
  - Klinikverbund Allgäu gGmbH ( Site 1408), Kempten (Allgäu), Bavaria
  - UKGM Gießen/Marburg ( Site 1404), Giessen, Hesse
  - Pius Hospital Oldenburg ( Site 1407), Oldenburg, Lower Saxony
  - St.-Antonius-Hospital ( Site 1411), Eschweiler, North Rhine-Westphalia
  - Universitätsklinikum Münster - Albert Schweitzer Campus ( Site 1405), Münster, North Rhine-Westphalia
  - Marienhaus Klinikum Mainz ( Site 1403), Mainz, Rhineland-Palatinate
- Greece (8):
  - UNIVERSITY HOSPITAL OF PATRAS-DIVISION OF ONCOLOGY ( Site 1452), Pátrai, Achaia
  - Errikos Dunant Hospital Center ( Site 1457), Athens, Attica
  - THORACIC GENERAL HOSPITAL OF ATHENS "I SOTIRIA"-3rd Dept of Internal Medicine and Laboratory, Oncol ( Site 1451), Athens, Attica
  - Metropolitan Hospital ( Site 1459), Athens, Attica
  - ATTIKON GENERAL UNIVERSITY HOSPITAL ( Site 1460), Chaïdári, Attica
  - University General Hospital of Herakleion ( Site 1458), Heraklion, Irakleio
  - University General Hospital of Larissa-Oncology Clinic ( Site 1453), Larissa, Thessaly
  - Papageorgiou General Hospital of Thessaloniki ( Site 1454), Thessaloniki
- Hungary (7):
  - Fejér Megyei Szent György Egyetemi Oktató Kórház ( Site 1506), Székesfehérvár, Fejér
  - Petz Aladár Megyei Oktató Kórház ( Site 1502), Győr, Győr-Moson-Sopron
  - Debreceni Egyetem Altalanos Orvostudomanyi Kar Tudogyogyaszati Tanszek ( Site 1508), Debrecen, Hajdú-Bihar
  - Mátrai Gyógyintézet ( Site 1504), Mátraháza, Heves County
  - Reformatus Pulmonologiai Centrum-Onkopulmonologiai Jarobeteg Centrum ( Site 1505), Törökbálint, Pest County
  - Somogy Vármegyei Kaposi Mór Oktató Kórház-Oncology center ( Site 1507), Kaposvár, Somogy County
  - Orszagos Koranyi Pulmonologiai Intezet ( Site 1501), Budapest
- Ireland (3):
  - Cork University Hospital ( Site 1553), Cork
  - St. James's Hospital ( Site 1554), Dublin
  - Tallaght University Hospital ( Site 1551), Dublin
- Israel (5):
  - Rambam Health Care Campus ( Site 1603), Haifa
  - Shaare Zedek Medical Center ( Site 1601), Jerusalem
  - Hadassah Medical Center ( Site 1605), Jerusalem
  - Meir Medical Center ( Site 1606), Kfar Saba
  - Sheba Medical Center ( Site 1602), Ramat Gan
- Italy (10):
  - AOU Renato Dulbecco ( Site 1661), Catanzaro, Calabria
  - Ospedale Santa Maria delle Croci ( Site 1652), Ravenna, Emilia-Romagna
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore ( Site 1653), Rome, Lazio
  - Fondazione Policlinico Universitario Campus Bio-Medico ( Site 1660), Rome, Roma
  - Istituto Nazionale Tumori Regina Elena ( Site 1651), Rome, Roma
  - Fondazione IRCCS Istituto Nazionale dei Tumori ( Site 1656), Milan
  - IEO Istituto Europeo di Oncologia ( Site 1655), Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 1657), Napoli
  - IRCCS Istituto Oncologico Veneto ( Site 1654), Padua
  - Centro Ricerche Cliniche di Verona ( Site 1659), Verona
- Japan (15):
  - Hospital of the University of Occupational and Environmental Health, Japan ( Site 1166), Kitakyushu, Fukuoka
  - St. Marianna University Hospital ( Site 1159), Kawasaki, Kanagawa
  - Kanagawa Cancer Center ( Site 1158), Yokohama, Kanagawa
  - Kindai University Hospital ( Site 1162), Sakai, Osaka
  - Shizuoka Cancer Center ( Site 1160), Sunto-gun, Shizuoka
  - Dokkyo Medical University Hospital ( Site 1152), Shimotsuga-gun, Tochigi
  - National Cancer Center Hospital ( Site 1156), Chūō, Tokyo
  - Tokyo Medical University Hospital ( Site 1157), Shinjuku, Tokyo
  - Chiba University Hospital ( Site 1154), Chiba
  - National Hospital Organization Kyushu Cancer Center ( Site 1167), Fukuoka
  - Fukushima Medical University Hospital ( Site 1151), Fukushima
  - Hiroshima University Hospital ( Site 1165), Hiroshima
  - Okayama University Hospital ( Site 1164), Okayama
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute ( Site 1161), Osaka
  - Wakayama Medical University Hospital ( Site 1163), Wakayama
- Netherlands (4):
  - Radboudumc ( Site 1706), Nijmegen, Gelderland
  - Maastricht UMC+ ( Site 1705), Maastricht, Limburg
  - Jeroen Bosch Hospital ( Site 1701), 's-Hertogenbosch, North Brabant
  - Medisch Centrum Leeuwarden ( Site 1702), Leeuwarden, Provincie Friesland
- New Zealand (3):
  - Tauranga Hospital-Bay of Plenty Clinical Trials Unit ( Site 2201), Tauranga, Bay of Plenty
  - Dunedin Hospital ( Site 2202), Dunedin, Otago
  - Waikato Hospital ( Site 2204), Hamilton, Waikato Region
- Peru (3):
  - Aliada ( Site 2753), Lima
  - Clínica Internacional - Sede San Borja ( Site 2752), Lima
  - Detecta Clínica ( Site 2751), Lima
- Poland (7):
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii ( Site 1763), Poznan, Greater Poland Voivodeship
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II ( Site 1756), Krakow, Lesser Poland Voivodeship
  - Instytut Gruźlicy i Chorób Płuc w Warszawie ( Site 1764), Warsaw, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu ( Site 1759), Przemyśl, Podkarpackie Voivodeship
  - Uniwersyteckie Centrum Kliniczne ( Site 1758), Gdansk, Pomeranian Voivodeship
  - Warmińsko - Mazurskie Centrum Chorób Płuc w Olsztynie ( Site 1760), Olsztyn, Warmian-Masurian Voivodeship
  - Swietokrzyskie Centrum Onkologii. ( Site 1754), Kielce, Świętokrzyskie Voivodeship
- Romania (3):
  - Centrul Medical Medicover Victoria ( Site 1802), Bucharest, București
  - Cabinet Medical Oncomed ( Site 1803), Timișoara, Timiș County
  - Institutul Regional de Oncologie ( Site 1804), Iași
- Singapore (2):
  - National Cancer Centre Singapore ( Site 2251), Singapore, Central Singapore
  - Tan Tock Seng Hospital ( Site 2252), Singapore, Central Singapore
- South Korea (7):
  - National Cancer Center ( Site 2305), Goyang-si, Kyonggi-do
  - The Catholic University of Korea St. Vincent s Hospital ( Site 2301), Suwon, Kyonggi-do
  - Ajou University Hospital ( Site 2306), Suwon, Kyonggi-do
  - Seoul National University Hospital ( Site 2303), Seoul
  - Severance Hospital Yonsei University Health System ( Site 2302), Seoul
  - Samsung Medical Center ( Site 2304), Seoul
  - Seoul St. Mary's Hospital ( Site 2307), Seoul
- Spain (7):
  - Hospital Insular de Gran Canaria ( Site 1911), Canarias, Canary Islands
  - Hospital Clinic de Barcelona ( Site 1919), Barcelona, Catalonia
  - Complejo Hospitalario Universitario A Coruna ( Site 1916), A Coruña, La Coruna
  - Hospital Universitario Quiron Madrid ( Site 1913), Pozuelo de Alarcón, Madrid
  - Hospital Universitari Vall D Hebron ( Site 1910), Barcelona
  - Hospital General Universitario Gregorio Maranon ( Site 1912), Madrid
  - Hospital Quiron Malaga ( Site 1914), Málaga
- Karolinska Universitetssjukhuset Solna ( Site 1951), Stockholm, Stockholm County, Sweden
- Taiwan (9):
  - Chung Shan Medical University Hospital ( Site 2351), Taichung
  - China Medical University Hospital ( Site 2358), Taichung
  - National Cheng Kung University Hospital ( Site 2354), Tainan
  - National Taiwan University Cancer Center (NTUCC) ( Site 2360), Taipei
  - Mackay Memorial Hospital ( Site 2355), Taipei
  - Taipei Medical University Hospital ( Site 2352), Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center ( Site 2359), Taipei
  - Taipei Veterans General Hospital ( Site 2357), Taipei
  - Chang Gung Memorial Hospital ( Site 2361), Taoyuan District
- Thailand (3):
  - Ramathibodi Hospital ( Site 2405), Ratchathewi, Bangkok
  - Faculty of Medicine - Khon Kaen University ( Site 2401), Muang, Changwat Khon Kaen
  - Maharaj Nakorn Chiang Mai Hospital ( Site 2404), Muang, Chiang Mai
- Turkey (Türkiye) (6):
  - Hacettepe Universite Hastaneleri ( Site 2001), Sıhhiye, Ankara
  - Sakarya Universitesi Tip Fakultesi Hastanesi ( Site 2006), Adapazarı, Sakarya
  - Namık Kemal University Medical Faculty ( Site 2007), Tekirdağ, Tekirdas
  - Ankara Bilkent Sehir Hastanesi ( Site 2002), Ankara
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi ( Site 2003), Istanbul
  - Karadeniz Technical University ( Site 2008), Trabzon
- United Kingdom (12):
  - Bristol Haematology and Oncology Centre ( Site 2072), Bristol, Bristol, City of
  - ROYAL MARSDEN HOSPITAL (CHELSEA)-Lung Unit ( Site 2075), London, Kensington and Chelsea
  - St Bartholomews Hospital ( Site 2052), London, London, City of
  - Royal Free Hospital ( Site 2074), London, London, City of
  - Guys Hospital ( Site 2057), London, London, City of
  - Royal Marsden Hospital (Sutton) ( Site 2076), London, London, City of
  - Nottingham City Hospital ( Site 2058), Nottingham, Nottinghamshire
  - St James University Hospital ( Site 2055), Leeds
  - Leicester Royal Infirmary ( Site 2051), Leicester
  - The Christie NHS Foundation Trust ( Site 2066), Manchester
  - The Clatterbridge Cancer Centre ( Site 2069), Metropolitan Borough of Wirral
  - Queen Alexandra Hospital ( Site 2059), Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26328&tenant=MT_MSD_9011